CLINICAL TRIAL: NCT02584387
Title: 3D Video Virtual Reality Exposure Therapy (3D-VVRET) Study
Brief Title: 3D Video Virtual Reality Exposure Therapy Study
Acronym: 3D-VVRET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Mark B. Powers, Research Associate Professor, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-08-0008
Record Dates: First submitted 2015-10-20; First posted 2015-10-22 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Acrophobia; Arachnophobia
MeSH Terms: conditions — Acrophobia; Arachnophobia

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- 3D VVRET (Experimental): Behavioral: 3D Video Virtual Reality Exposure Therapy (VVRET)
  1 30 minute 3D VRET treatment session for arachnophobia.
  Interventions: Behavioral: 3D Video Virtual Reality Exposure Therapy
- Waitlist (No Intervention): Participants randomized to the waitlist group will complete all study procedures except the 3D VVRET. After the conclusion of their sessions, these participants will be offered the full 3D-VVRET treatment.

INTERVENTIONS:
Behavioral: 3D Video Virtual Reality Exposure Therapy — The 3D video exposure therapy treatment will be administered using an oculus rift virtual reality headset. The oculus rift is a new, affordable virtual reality headset, which uses two different spherical lenses to induce a sense of stereoscopic 3D. Ortho-stereoscopic 3D refers to 3D videos that are designed to mimic the natural depth we normally see, as opposed to exaggerating it (i.e. Commercial 3D movies). To create these 3D videos, the UT 3D Department shot videos of live spiders using a stereoscopic 3D dual camera rig, which simultaneously shoots footage with two cameras positioned apart from each other in a way that mimics the natural pupillary distance between our right and left eyes. To create a sense of 3D depth, the footage of the right and left cameras is then projected on the two different lenses of the oculus rift, creating a sense of depth to the viewer through retinal disparity.
  Arms: 3D VVRET

SUMMARY:
This study seeks to examine a Virtual Reality Exposure Therapy (VRET) using the 3D Video Virtual Reality (VR) technology for the fear of spiders.

DETAILED DESCRIPTION:
An estimated 10-11% of the US population experiences a specific phobia at some point in their lives (American Psychiatric Association, 1994; Magee et al., 1996). About 60-85% of those individuals with a specific phobia never seek treatment (Agras, Sylvester, & Oliveau, 1969; Boyd et al., 1990; Magee et al., 1996). Clinical psychologist can help improve the number of phobia sufferers to seek treatment. Advances in technology are helping clinicians create novel treatment strategies for different anxiety disorders. Virtual reality exposure therapy (VRET) may help these individuals confront their fears and treat their phobia.

While virtual reality exposure therapy has shown promise in research (Powers & Emmelkamp, 2008), studies have shown that many users complain that the computer generated virtual reality (VR) stimuli looks unrealistic, eccentric and too much like a video game (Kwon, Powell, & Chalmers, 2013). Virtual reality environments have been traditionally created by programmers using video game assets and computer generated imagery (CGI). While CGI can be used to make intricate virtual environments, unless there is a team of expert digital artists, the virtual stimulus may end up looking rudimentary and exhibit a number of graphical glitches which could prove distracting in therapy. Furthermore CGI often suffers from the uncanny valley effect: the tendency of CGI representations of people to be viewed as unsettling as the representations become more lifelike. In addition the many current CGI virtual reality packages are expensive and only available for limited number of fear domains. Recently however an exciting alternative to traditional computer generated virtual reality has emerged: ortho-stereoscopic 3D Video VR. Ortho-stereoscopic 3D refers to 3D videos that are designed to mimic the natural depth we normally see, as opposed to exaggerating it (i.e. Commercial 3D movies). The benefit of 3D VR as opposed to CGI VR is that it is photo realistic, does not suffer from a uncanny valley effect of CGI, and is able to capture nuances of real life fears that are hard to reproduce with CGI.

ELIGIBILITY:
Inclusion Criteria:

* • Between the ages of 18 and 65

  * At least one standard deviation above the SONA pool mean on Fear of Spiders Questionnaire or Acrophobia Questionnaire.

Exclusion Criteria:

* • Hearing or visually impaired where they cannot use the VRET gear

  * Currently (or in the last 3 months) receiving exposure-based treatment for acrophobia or arachnophobia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-09; Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Fear of Spiders Questionnaire | Pre-treatment and 1 week follow-up

SECONDARY OUTCOMES:
Behavioral Approach Test | Pre-treatment and Post-treatment
Acceptance and Action Questionnaire | Pre-treatment
State-Trait Anxiety Inventory | Pre-treatment
Anxiety Sensitivity Index (ASI-3) | Pre-treatment
Distress Tolerance Scale (DTS) | Pre-treatment
Disgust Emotion Scale | Pre-treatment
Disgust Propensity and Sensitivity Scale (DPSS-R) | Pre-treatment

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Texas at Austin, Austin, Texas, United States